CLINICAL TRIAL: NCT02708641
Title: A Phase II Study of Pembrolizumab as Post-Remission Treatment of Patients ≥ 60 With Acute Myeloid Leukemia (AML) Who Are Not Transplantation Candidates
Brief Title: A Phase II Study of Pembrolizumab as Post-Remission Treatment of Patients ≥ 60 With AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Boyiadzis (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Michael Boyiadzis, Associate Professor of Medicine, Division of Hematology Oncology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-101
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AML patients (Experimental): pembrolizumab 200 mg given IV once every three weeks
  Interventions: Drug: pembrolizumab

INTERVENTIONS:
Drug: pembrolizumab — 200 mg IV given every three weeks
  Other Names: Keytruda

SUMMARY:
This study evaluates the effect of pembrolizumab on the duration of remission in acute myeloid leukemia. Pembrolizumab is given after complete remission is obtained in those with AML at least 60 years old who are not candidates for allogeneic stem cell transplant. The primary purpose of this study is determine if the time to relapse can be extended. Additionally, the safety and tolerability of pembrolizumab will be closely monitored.

DETAILED DESCRIPTION:
Patients >60 years old with AML often have a dismal prognosis. Even though many of these patients are able to obtain a Complete Response to treatment, relapse occurs in the vast majority of patients. Transplants may reduce relapse rates in this population, but is only feasible in a minority of patients. AML's immunosuppressive microenvironment in general and PD-1/PD-L1 upregulation in particular appears to increase the risk of relapse. Importantly, PD-1 and its ligands are particularly increased after therapy compared to initial diagnosis. As such, PD-1 inhibition with pembrolizumab offers to limit leukemic cell immune escape, thereby allowing the patient's immune system to eradicate the submicroscopic residual disease and reducing relapse rates.

Treatment for this study is 200 mg Q3W as an appropriate dose for the switch to fixed dosing is based on simulations performed using the population PK model of Pembrolizumab showing that the fixed dose of 200 mg every 3 weeks will provide exposures that 1) are optimally consistent with those obtained with the 2 mg/kg dose every 3 weeks, 2) will maintain individual patient exposures in the exposure range established in melanoma as associated with maximal efficacy response and 3) will maintain individual patients exposure in the exposure range established in melanoma that are well tolerated and safe.

ELIGIBILITY:
Inclusion Criteria:

* be willing and able to provide written informed consent for the trial
* be ≥ 60 years of age on day of signing informed consent
* have a newly diagnosed AML based on the World Health Organization (WHO) criteria, currently in first complete remission (CR) on a bone marrow biopsy performed within 4 weeks of treatment initiation
* have received the last dose of induction or consolidation chemotherapy within 3 months of treatment initiation
* not be eligible for or willing to proceed with allogeneic stem cell transplant or for whom allogeneic stem cell transplant is not considered standard of care
* have a performance status of ≤ 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* demonstrate adequate organ function, with all screening labs performed within 10 days of treatment initiation
* transfusion independent (no red blood cell or platelet transfusions in the preceding 2 weeks of screening)
* negative urine and/or serum pregnancy test
* subjects of reproductive potential must agree to use acceptable birth control method

Exclusion Criteria:

* have a diagnosis of Acute Promyelocytic Leukemia (APL) as defined by the WHO
* currently participating in or has participated in a study of an investigational agent or device within 4 weeks of treatment initiation
* have a diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to treatment initiation
* have prior monoclonal antibody within 4 weeks prior to study Day 1 or have not recovered from adverse events due to agents administered more than 4 weeks earlier
* have prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 have not recovered from adverse events due to previously administered agent(s)
* have a known additional malignancy that is progressing or requires active treatment except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* have known active central nervous system (CNS) involvement
* have an active autoimmune disease requiring systemic treatment within the past 3 months
* has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* have an uncontrolled, life-threatening active infection
* have a history or current evidence of condition, therapy, or laboratory abnormality that would preclude study participation in the opinion of the treating investigator
* have known psychiatric or substance abuse disorders that would interfere with cooperation with the trial requirements
* is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial
* have received prior therapy with any antibody targeting the T-cell co-stimulation or checkpoint pathways
* have a known history of HIV
* have known active Hepatitis B or Hepatitis C
* have received a live vaccine within 30 days prior to treatment initiation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boyiadzis, MD, MHSc, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembro 200 mg - AML Patients: Patients with AML (not transplantation eligible) treated with pembrolizumab 200 mg IV administered once every three weeks, post-remission
Period: Overall Study
Arm/Group | Pembro 200 mg - AML Patients
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembro 200 mg - AML Patients
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 70.4 [60.2 to 82.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
ECOG Performance Status [Count of Participants; unit: Participants] — The ECOG Performance Status is a measure of functional status used as a selection criterion for cancer research. Scores range from 0 to 5. Scoring information: 0 = Fully active; no performance restrictions; 1 = Strenuous physical activity restricted; fully ambulatory and able to carry out light work; 2 = Capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours; 3 = Capable of only limited self-care; confined to bed or chair >50% of waking hours; 4 = Completely disabled; cannot carry out any self-care; totally confined to bed or chair.
  Participants
    ECOG = 0 | 4
    ECOG = 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse (TTR)
Description: Time to recurrence of AML, including only deaths related to recurrence. Relapse of AML is defined as patients reaching remission (bone marrow contains <5% blast cells, blood cell counts return to within normal limits, no signs disease) followed by a return of leukemia cells in the marrow and a decrease in normal blood cells.
Time Frame: Up to 24 months
Population: Patients who received at least one cycle of study treatment and were evaluable for response.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Pembro 200 mg - AML Patients
Number analyzed (Participants) | 12
months | 12.14 [9.00 to NA] — Upper bound of CI not reached (due to low accrual number)

2. Primary Outcome: Worst Grade of Adverse Events Experienced (Unrelated to Relatedness to Study Therapy)
Description: Worst Grade of AE experienced, regardless of relatedness to study therapy, per CTCAE v5.0.
Time Frame: Up to 24 months
Population: Patients who received at least one cycle of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembro 200 mg - AML Patients
Number analyzed (Participants) | 12
Participants
  Grade 2 | 1
  Grade 3 | 6
  Grade 4 | 5

3. Primary Outcome: Worst Grade of Adverse Events Experienced (at Least Probably Related to Treatment)
Description: Worst Grade of AE experienced, at least probably related to treatment, per CTCAE v5.0.
Time Frame: Up to 24 months
Population: Patients who received at least one cycle of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembro 200 mg - AML Patients
Number analyzed (Participants) | 12
Participants
  Grade 2 | 3
  Grade 3 | 5
  Grade 4 | 4

4. Primary Outcome: Worst Grade of Adverse Events Experienced (at Least Probably Related to Treatment)
Description: Worst Grade of AE experienced, at least probably related to treatment, per CTCAE v5.0.
Time Frame: Up to 24 months
Population: Patients who received at least one cycle of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembro 200 mg - AML Patients
Number analyzed (Participants) | 12
Participants
  Grade 1 | 3
  Grade 2 | 1
  Grade 3 | 1
  Grade 4 | 1

5. Secondary Outcome: Overall Survival (OS)
Description: The length of time from date of start of treatment that patients are still alive.
Time Frame: Up to 48 months
Population: Patients eligible for study participation.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Pembro 200 mg - AML Patients
Number analyzed (Participants) | 12
months | 42.18 [14.65 to NA] — Upper bound of CI not reached (due to low accrual number)

6. Other Pre Specified Outcome: Quantification of Activated T Cells
Description: Determination of activated T cells level (percentages) in peripheral blood. Increased levels of activated T cells may indicate decreasing disease progression.
Time Frame: Up to 24 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Quantification of Activated NK Cells
Description: Determination of activated NK cells level (percentages) in peripheral blood. Increased levels of activated T cells may indicate decreasing disease progression.
Time Frame: Up to 24 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Quantification of Regulatory T Cells (Treg)
Description: Determination of regulatory T cell (Treg) levels (percentages) in peripheral blood. Treg cells are involved in cancer progression by inhibiting anti-cancer immunity. Increased levels of Treg cells may indicate progressing disease.
Time Frame: Up to 24 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Cytokine Expression
Description: Determination of cytokine expression levels (percentages) in peripheral blood. Cytokine expression is associated with cancer progression, immuno-suppression, and decreased anti-cancer response.
Time Frame: Up to 24 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Granzyme B/Perforin Expression
Description: Determination of Granzyme B/perforin expression levels (percentages) in peripheral blood.
  Granzyme B/perforin expression is associated with the suppression of cancer progression.
Time Frame: Up to 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events monitored up to 24 months, All-Cause Mortality monitored up to 48 months
Description: Adverse Events: Grade 1 and Grade 2 events per CTCAE v4.0 Serious Adverse Events: Grade 3 and Grade 4 events per CTCAE v4.0
Arm/Group | AML Patients
All-Cause Mortality (participants affected / at risk) | 6/12
Serious Adverse Events (participants affected / at risk) | 11/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AML Patients (N=12)
Anemia (Blood and lymphatic system disorders) | 2
Blood and lymphatic system (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 2
Colitis (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
General disorders and admin. site (General disorders) | 1
Appendicitis (Infections and infestations) | 1
Infections and infestations (Infections and infestations) | 1
Lung infection (Infections and infestations) | 3
Rhinitis infective (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 6
Platelet count decreased (Investigations) | 6
White blood cell decreased (Investigations) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hematuria (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AML Patients (N=12)
Acute coronary syndrome (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Floaters (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Lung infection (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Scrotal infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Cholesterol high (Investigations) | 1
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition (Metabolism and nutrition disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hemoglobinuria (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Scrotal pain (Reproductive system and breast disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Infections and infestations (Infections and infestations) | 2
Vaginal infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 2
Act. partial thrombop. time prolonged (Investigations) | 2
INR increased (Investigations) | 2
Investigations - Other, specify (Investigations) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Cardiac disorders - Other, specify (Cardiac disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 3
General disorders and admin. site (General disorders) | 3
Creatinine increased (Investigations) | 3
Neutrophil count decreased (Investigations) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Musculoskeletal and connective tissue (Musculoskeletal and connective tissue disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Skin and subcut. tissue (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 3
Edema limbs (General disorders) | 4
Pain (General disorders) | 4
Lymphocyte count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Sinus tachycardia (Cardiac disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 5
Fever (General disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 6
Anemia (Blood and lymphatic system disorders) | 7
Fatigue (General disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT02708641/Prot_SAP_000.pdf